CLINICAL TRIAL: NCT03774290
Title: A Phase II, Double-blind, Randomized, Parallel-group, Placebo- Controlled Multi-center Study to Investigate the Effect of the Adenosine A1 Receptor Antagonist PBF-680 on Forced Expiratory Volume in 1 Second (FEV1) in Patients With Mild-to-moderate Persistent Atopic Asthma
Brief Title: Study to Investigate the Effect of PBF-680 on Forced Expiratory Volume in 1 Second (FEV1) in Asthmatic Patients
Acronym: ADENOASMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Pivotal S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBF-680CT-05
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBF-680 10 mg (Experimental): 10 mg of PBF-680 once a day
  Interventions: Drug: PBF-680
- Placebo oral capsules (Placebo Comparator): Placebo once a day
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: PBF-680 — PBF-680 is an adenosine A1 receptor antagonist
  Arms: PBF-680 10 mg
Drug: Placebo oral capsule — Oral gelatine capsule
  Arms: Placebo oral capsules

SUMMARY:
The present trial is an exploratory study aiming at evaluating the safety, tolerability, and efficacy of a 15-day, once daily administration of 10 mg PBF-680 in subjects with persistent, mild-to-moderate atopic asthma.

DETAILED DESCRIPTION:
Purpose and rationale: Extracellular adenosine, produced from dephosphorylation of adenosine triphosphate (ATP) and adenosine monophasphate (AMP), is an important signaling molecule in asthma, involved in bronchoconstriction and airway inflammation. PBF-680 is an A1 adenosine receptor antagonist that has successfully completed single dose escalation and treatment-period phase-I trials in healthy volunteers, plus a crossover, proof-of-concept Phase-IIa trial in mild and moderate asthmatics, where a single dose significantly attenuated airway hyperresponsiveness to AMP challenge and increased 8-hour post-challenge FEV1. In terms of exploratory efficacy, the primary purpose of this study is to determine whether PBF-680 compared to placebo, improves the FEV1, as well as to provide comparative safety data from this population of asthmatics. Measurements made in this study will also be used to establish whether this treatment improves other variables related to asthma control and lung function.

Objectives: The primary objective is to demonstrate an improvement in trough FEV1 upon a 15-day treatment with PBF-680 compared to placebo in mild-to-moderate asthmatics that, on study entry, are managed in Global Initiative for Asthma (GINA) therapeutic steps 2-3. Secondary objectives include determinations of FEV1 area under the curve (AUC), evaluations on pre- and post- bronchodilator FEV1, and patient reported outcomes (PROs) including Asthma Control Questionnaire-7 (ACQ-7) and Standardized Asthma Quality of Life Questionnaire (AQLQ(S)).

Study design and population: this is a multicenter, double-blind, randomized, placebo- controlled trial with a 2-arm parallel design. The treatments studied are once-daily PBF- 680 10 mg and placebo, as two orally administered, 5-mg PBF-680 capsules or two placebo capsules, respectively. The study comprises: (i) a minimum of 5-days screening period, during which, the subject's clinical stability and overall eligibility for the study will be assessed; (ii) a weaning phase where a stepwise tapering of the asthma medication will be done upon 7-day periods; (iii) the randomized, parallel-arm treatment period; and (iv) an end-of-study follow-up visit. The asthma medication weaning period comprises three possible visit pathways in order to adjust for each subject's asthma therapy on study entry. The study will comprise a primary analysis population of 58 stable asthmatic subjects managed as described for the objectives, who meet all inclusion criteria and no exclusion criteria and complete a full, valid data set for the primary variable. The total recruitment estimates to meet this target is 78 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any study assessments are performed. Subjects must be able to communicate well with the investigator and staﬀ so that they can understand and comply with the requirements of the study.
* Male and female subjects of 18-65 years age.
* Subjects with a medical history of mild-to-moderate persistent allergic asthma, diagnosed according to GINA 2017 guidelines, and managed in therapeutic steps 2-3 being inhaled corticosteroid (ICS) limited to low/medium dose, or step 4 restricted to medium-dose ICS plus ong-acting beta2-agonist (LABA) and/or a leukotriene antagonist, as maintenance therapy.
* A positive skin prick test to aeroallergens, such as house dust mite, tree or grass pollen, pet dander, or cockroach antigens. In addition, any allergens speciﬁc to the country/locality can be included.
* Women of child-bearing potential must agree to employ eﬀective contraception from Visit 1 through FU visit, unless they are surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), are at least 2 years postmenopausal, or practice abstinence.
* All female subjects must have negative pregnancy test results at screening and baseline.
* Male subjects must agree to use two acceptable methods of contraception, (e.g. spermicidal gel plus condom) for the entire duration of the study and up to the study completion visit, and refrain from fathering a child within the three months following the last study drug administration. Periodic abstinence and withdrawal are not acceptable methods of contraception.
* Subjects must weigh at least 45 kg and must have a body mass index (BMI) ≥ 17 kg/m2.
* Evidence of asthma as documented by either:

Subjects must demonstrate an increase of ≥12% AND ≥200 mL in FEV1 over their pre- bronchodilator value within 30 min after inhaling a total of 400 μg of salbutamol (reversibility test). Reversibility can be documented prior to Screening (Visit 1) or determined at screening or during the weaning period up to visit V5.

Or documented history of bronchial hyper reactivity (e.g. fall in FEV1 from baseline of more than or equal to 20 percent with inhaled standard doses of Adenosine monophosphate, methacholine or histamine, or more than or equal to 15 percent with standardized hyperventilation, hypertonic saline or mannitol challenge) from a bronchoprovocation study [e.g. methacholine challenge prior to Screening (Visit 1)].

Or a decrease ≥ 5% of their initial FEV1 measured at V1 during the weaning period up to visit V5.

* Subjects must have either a pre-bronchodilator FEV1 ≥60% and ≤90% of their predicted normal value upon completion of LABA and ICS weaning on Visit 5 or a decrease ≥ 5% of their initial FEV1 measured at V1 during the weaning period up to visit V5.
* Subjects must have an ACQ-7 score ≥1.5 upon completion of LABA and ICS weaning on Visit 5.
* Subjects must meet a ≥80% compliance with the morning and evening electronic/PEF meter recordings during the weaning of their asthma maintenance therapy (i.e. from visit V2 to visit V5).

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* History of hypersensitivity to the study medication or drugs of similar chemical classes (A1 adenosine receptor antagonists).
* A history of clinically signiﬁcant ECG abnormalities or a recent history of autonomic dysfunction (e.g. recurrent episodes of fainting, arrhythmia, etc.).
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
* Pregnant or nursing (lactating) women.
* Smokers, deﬁned by smoking within the previous 6 months or having a smoking history of more than 10 packs-years, a pack-year being deﬁned as smoking the equivalent of 20 cigarettes (a pack) per day for 1 year.
* Subjects with severe persistent asthma managed in GINA therapeutic step 4 (except for the restricted allowance in inclusion criterion 3) or 5 according to GINA 2017 guidelines. This criterion includes subjects treated with high-dose ICS, systemic corticosteroids, tiotropium bromide, theophylline or monoclonal antibody-based biological therapies such as omalizumab, mepolizumab, reslizumab, etc. Subjects treated with any immunosuppressant drug, or with systemic corticosteroids for any condition other than asthma, are excluded. Subjects requiring daily use of antihistamine drugs are also excluded.
* Present or past use of a biologic (e.g. monoclonal antibodies) agent for the treatment of asthma. Use of a biologic agent for any other condition within the past 6 months.
* Use of systemic corticosteroids to treat an asthma exacerbation or any other condition within 4 weeks prior to Visit 1.
* History of life-threatening asthma, deﬁned as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest and/or hypoxic seizures. History of asthma exacerbations that required ward hospitalization or an emergency room stay greater than 48 hours within 5 years prior to Visit 1.
* Any disease or illness other than asthma that may require the use of systemic corticosteroids during the study period.
* Any occupational exposure to allergens/irritants that may have a potential to worsen the asthma symptoms during the trial.
* A respiratory tract infection requiring the use of antibiotics within 4 weeks prior to visit V1, or pneumonia within 6 months prior to visit V1.
* An asthma exacerbation requiring treatment or the use of any health care resources within 4 weeks prior to visit V1. This includes asthma exacerbations managed with a transient increase of the subject's regular asthma maintenance therapy, and self- managed exacerbations using an "action plan".
* Subjects with any other underlying diseases that may compromise safety or may interfere with eﬃcacy outcomes (e.g. tuberculosis, clinically relevant bronchiectasis, diﬀuse lung interstitial disease, pulmonary hypertension, emphysema, chronic bronchitis, alpha-1-antitrypsin deﬁciency, systemic immune-driven disorders).
* The use of prescription or over-the-counter medications is subjected to protocol- established restrictions (non-permitted medications)
* Any surgical or medical condition which might signiﬁcantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The investigator must determine this in consideration of the subject's medical history and/or clinical or laboratory evidence of the following conditions, including but not limited to: inﬂammatory bowel disease; digestive tract ulcers; gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy or bowel resection; pancreatic injury or pancreatitis; liver disease or liver injury as indicated by abnormal liver function.
* Subjects that are receiving, or have received within the past 5 years, speciﬁc immunotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Effect of PBF-680 on trough forced expiratory volume in 1 second (FEV1) | 16 Days
  Defined as the average of the FEV1 measurements taken at 23h 15min and 23h 45min post-dose after the final dose.

SECONDARY OUTCOMES:
Effect of PBF-680 in the FEV1 area under curve AUC30min-23h 30min post-dose | 16 days
  Defined as the FEV1 area under curve of a serial of spirometries from 30min-23h 30min post-dose through days 15-to-16
Effect of PBF-680 in the standardized FEV1 AUC30min-6h post- dose | 15 Days
  Defined as the FEV1 area under curve of a serial of spirometries from 30min-6h post-dose on day 15
Effect of PBF-680 in the pre-bronchodilator FEV1 | 8 days
  Defined as the FEV1 before use of bronchodilator at pre-dose spirometry on day 8
Effect of PBF-680 in the post- bronchodilator FEV1 at pre-dose spirometry on day 8 | Day 8 and Day 16
  Defined as the FEV1 after use of bronchodilator at pre-dose spirometry on day 8 and 16
Effect of PBF-680 on the asthma control as measured by Asthma Questionnaires | Day 8 and Day 15
  Asthma Control Questionnaire (ACQ-7) comprises 5 patient-reported symptoms that are scored from 0 to 6.The points are added and divided by 5. According to the result:
  Less than or equal to 0.75: Adequate control of asthma From 0.75 to 1.50: partially controlled asthma More than 1.50: Inadequate control of asthma. The Asthma Quality of Life Questionnaire AQLQ(S) scores symptoms, activity limitation, emotional function, and environmental exposure through 32 questions. The overall AQLQ score is the mean of the responses to each-of the 32 questions on a 7- point scale (7=no impairment, 1 =severe impairment)
Effect of PBF-680 on daily, morning and evening FEV1 and PEF as measured by an electronic diary/Peak Expiratory Flow (PEF) meter device. | 16 days
  On each morning and evening, the subjects must ﬁll the diary questions and record three brief expiratory maneuvers that generate PEF and FEV1 data.
Effect of PBF-680 in the use of rescue bronchodilator as reported by the subject using an electronic diary/PEF meter device. | 16 days
  On each morning and evening, the subjects must ﬁll the diary questions and record three brief expiratory maneuvers that generate PEF and FEV1 data
Number of subjects with treatment-related adverse events as assessed by CTCAE v4 | 16 days
  Adverse events will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4

CONTACTS AND LOCATIONS:
Locations (1):
- Unitat de Pneumologia Experimental, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No